CLINICAL TRIAL: NCT01180205
Title: A TElmisartan and AMlodipine STudy to Assess the Cardiovascular PROTECTive Effects as Measured by Endothelial Dysfunction in Hypertensive at Risk Patients Beyond Blood Pressure
Brief Title: Telmisartan, Amlodipine and Flow Mediated Dilation
Acronym: TEAMSTAprotect
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Prof.Dr.med.S.Blankenberg, Departement for cardiology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009-017010-68
Record Dates: First submitted 2010-08-04; First posted 2010-08-12 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2010-04

CONDITIONS: Hypertension
Keywords: FMD; hypertension; Telmisartan; Amlodipine
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Amlodipine; Olmesartan Medoxomil; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- T/A (Active Comparator): Telmisartan + Amlopidpine
  Interventions: Drug: Telmisartan; Drug: Amlodipine
- O/HCT (Active Comparator): Olmesartan + Hydrochlorothiazide
  Interventions: Drug: Olmesartan medoxomil; Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Telmisartan — Telmisartan (80 mg ,Tablets, QD, p.o., 26 weeks)
  Other Names: MICARDIS® (Telmisartan)
  Arms: T/A
Drug: Amlodipine — Amlodpine 5 mg po 14 days, the forced - titration to 10 mg po for 24 weeks
  Other Names: Norvasc
  Arms: T/A
Drug: Olmesartan medoxomil — Olmesartan 40 mg po for 26 weeks
  Other Names: Olmetec
  Arms: O/HCT
Drug: Hydrochlorothiazide — HCT 12,5 mg po for 14 days, then 25 mg po for 24 weeks
  Arms: O/HCT

SUMMARY:
To show superior effects of the combination Telmisartan and Amlodipine (T and A) vs Olmesartan and Hydrochlorothiazide (O and HCTZ) on endothelial dysfunction as measured by flow mediated dilation (FMD) in hypertensive at risk patients beyond bloodpressure BP (equal BP in both arms; target BP <140/90 mmHg (<130/80 mmHg for renally impaired and/ or diabetic patients). To investigate the effects of T and A vs O and HCTZ in reducing arterial stiffness and carotid atherosclerotic plaques.

DETAILED DESCRIPTION:
This is a Phase IV, randomised, double-blind, forced- titration, active controlled, mono-center study to primarily compare the effects on endothelial function of the combination of telmisartan and amlodipine versus olmesartan and hydrochlorothiazide in hypertensive patients at risk beyond blood pressure. Additionally, key secondary endpoints for this trial are the changes in plaque and intima media complex echogenicity and the change in arterial stiffness after 26 weeks of treatment.

576 patients will be included in the study after a screening period of two weeks and then randomised in one of the two treatment groups. Pretreatment with ARBs, ACE-Inhibitors, amlodipine and diuretics will be stopped last day before visit 2. At visit 2 the treatment with either telmisartan and amlodipine or olmesartan and hydrochlorothiazide starts, so that no medication is stopped without having been replaced by the study medication. After two weeks treatment all patients will be up-titrated and having the maintenance dose for the following 24 weeks. The trial will be performed at one center in Germany with access to patients with hypertension. Patients will be recruited from the Department of Cardiology of the university Mainz. There will be a promotion flyer and an information booklet about the study for cardiologists practicising near Mainz, who like to sent their patient to the study center. Sponsor of the trial is the university Mainz.

Stefan Blankenberg, MD has been designated as Principal Investigator for this national, mono-center trial.

The study will be completed when the last patient had his last visit and the telephone follow - up two weeks later will be performed. This latest patient contact is defined as end of trial.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent in accordance with Good Clinical Practice and local legislation.
* Age 35 and older.
* Male and female, treated and treatment-naive patients with uncontrolled hypertension (defined as 20/10 mmHg above target BP of <140/90 mmHg [<130/80 mmHg for renally impaired and/ or diabetics patients])
* Male and female treated patients with controlled hypertension (defined as target BP < 140/90 mmHg [ < 130/80 mmHg for renally impaired and/ or diabetics patients])
* > 3 cardiovascular risk factors CVRFs and/or metabolic syndrome and/or diabetes mellitus and/or end organ damage

Exclusion Criteria:

1. Pretreatment with Telmisartan within the last 3 months.
2. Pretreatment with Amlodipine, Diuretics and AT1Blocker/ACEInhibitor within the last 3 months
3. Myocardial infarction within last 6 months.
4. Previous stroke or hemodynamically relevant stenosis of carotic arteria (>70%).
5. Previous cardial or peripheral bypass surgery within last 6 months.
6. PAD stadium III - IV n.F.
7. Chronic heart failure NYHA III- IV.
8. Unstable angina.
9. Known intolerance to angiotensin receptor blockers, diuretics or dihydropyridine calcium channel blocker.
10. Pre-menopausal women (last menstruation ≤1 year prior to signing informed consent) who:

    1. are not surgically sterile; or
    2. are nursing, or
    3. are pregnant, or
    4. are of childbearing potential and are NOT practicing acceptable methods of birth control, or do NOT plan to continue practicing an acceptable method throughout the trial.

       The only acceptable methods of birth control are:
    5. Intra-Uterine Device (IUD)
    6. Oral
    7. implantable or injectable contraceptives
    8. Estrogen patch
    9. Hormonal birth control should have been in use for at least three months before the study and continue at least until the next menstrual period after completing the study
11. Night shift workers who routinely sleep during the daytime and whose work hours include midnight to 4:00 a.m.
12. Known or suspected secondary hypertension (e.g., renal artery stenosis or phaeochromocytoma)
13. Mean in-clinic seated cuff SBP ≥180 mmHg and/or DBP ≥110 mmHg
14. Renal dysfunction as defined by the following laboratory parameters:
15. Serum creatinine >3.0 mg/dL (or >265 μmol/L) and/or known estimated creatinine clearance of <30 ml/min and/or clinical markers of severe renal impairment.
16. Bilateral renal artery stenosis, renal artery stenosis in a solitary kidney, post-renal transplant patients or patients with only one kidney
17. Clinically relevant hypokalemia or hyperkalemia (i.e., <3.0 or >5.5 mEq/L, may be rechecked for suspected error in result)
18. Uncorrected sodium or volume depletion
19. Primary aldosteronism
20. Hereditary fructose intolerance
21. Biliary obstructive disorders (e.g., cholestasis) or hepatic insufficiency
22. Clinically significant ventricular tachycardia, atrial fibrillation, atrial flutter or other clinically relevant cardiac arrhythmias as determined by the Investigator
23. Hypertrophic obstructive cardiomyopathy, severe obstructive coronary artery disease, aortic stenosis, hemodynamically relevant stenosis of the aortic or mitral valve
24. Patients whose diabetes has not been stable and controlled for at least the past three months as defined by an HbA1C ≥10%
25. Patients who have previously experienced symptoms characteristic of angioedema during treatment with ACE inhibitors or angiotensin-II receptor antagonists
26. History of drug or alcohol abuses within six months prior to signing the informed consent form
27. Concomitant administration of any medications known to affect BP, except medications allowed by the protocol
28. Any investigational drug therapy within one month of signing the informed consent
29. Known contraindication to any component of the trial drugs (telmisartan, amlodipine, olmesartan, hydrochlorothiazide)
30. History of non-compliance or inability to comply with prescribed medications or protocol procedures
31. Any other clinical condition which, in the opinion of the investigator, would not allow safe completion of the protocol and safe administration of the trial medication

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 576 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-10 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
FMD flow mediated dilation | baseline
  The overall mean improvement following 26 weeks of treatment in FMD as measured by the change from Visit 2 for T80/A10 is equal to O40/H25.
FMD | after 26 weeks
  The overall mean improvement following 26 weeks of treatment in FMD as measured by the change from Visit 2 for T80/A10 is equal to O40/H25.

SECONDARY OUTCOMES:
Echogenicity | baseline
  To investigate the effects of T and A vs O and HCTZ on grayscale median of carotid atherosclerotic plaques
arterial stiffness | baseline
  To investigate the effects of T and A vs O and HCTZ in reducing arterial stiffness
arterial stiffness | after 26 weeks
  To investigate the effects of T and A vs O and HCTZ in reducing arterial stiffness
Echogenicity | after 26 weeks
  To investigate the effects of T and A vs O and HCTZ on grayscale median of carotid atherosclerotic plaques

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Blankenberg, Prof.Dr.med., Principal Investigator — Universitätsmedizin Mainz, II.Medizinische Klinik
Locations (1):
- Universitätsmedizin Mainz, Mainz, Rhineland-Palatinate, Germany